CLINICAL TRIAL: NCT06535087
Title: The Impact of Airway Allergic Diseases on the Health-related Quality of Life of Children and Their Parents (Caregivers): A Prospective Controlled Study
Brief Title: The Impact of Airway Allergic Diseases on Children's and Parents' Quality of Life
Status: Recruiting | Type: Observational
Sponsor: Wenjing Zhou (Other)
Responsible Party: Sponsor-Investigator, Wenjing Zhou, Principal Investigator, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: IIT-2024-0110
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Asthma; Rhinitis, Allergic; Quality of Life
Keywords: pediatric allergic disease, health-related quality of life
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Alutard SQ allergen; Omalizumab; Budesonide; Terbutaline; montelukast; Cetirizine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — complete blood count
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Allergic disease group: Receiving: 1) Subcutaneous immunotherapy and 2) Standard Treatment for Asthma and Rhinitis.
  Interventions: Drug: Subcutaneous immunotherapy / Standard Treatment for Asthma and Rhinitis
- Healthy control Group: Healthy children aged 5-16 from the Shanghai region, with no history of allergic diseases, and without any intervention.

INTERVENTIONS:
Drug: Subcutaneous immunotherapy / Standard Treatment for Asthma and Rhinitis — 1. Subcutaneous Allergen-Specific Immunotherapy:
     * Pre-treatment: Omalizumab subcutaneous injection, with the total IgE level serving as the basis for calculating the dosage for children. The appropriate dosage of omalizumab (each dose ranging from 75 to 600 mg) and administration frequency (once every 4 weeks) are determined based on the baseline IgE (IU/mL, measured before the start of treatment) and body weight (kg).
     * Mite Allergen Preparation: (Antergen/Alutard)
  2. Standard Treatment:
     * Asthma: Inhaled corticosteroids (ICS) combined with long-acting beta-2 agonists, leukotriene receptor antagonists.
     * Allergic Rhinitis: Oral antihistamines, nasal antihistamines, nasal corticosteroids, anti-leukotriene drugs, cromolyn sodium, decongestants (oxymetazoline hydrochloride), and nasal saline irrigation.
  Other Names: Alutard; Antergen; Xolair; Pulmicort; Bricanyl; Singulair; Zyrtec
  Groups: Allergic disease group

SUMMARY:
This prospective observational study aims to assess the health-related quality of life (HRQoL) of 200 children (ages 5-16) with bronchial asthma, allergic rhinitis, or both, and their 200 parents, comparing 100 children receiving specific immunotherapy with 100 receiving routine treatment. Using EQ-5D-Y(EuroQol five dimensions questionnaire, youth version), disease-specific scales, and newly developed Chinese versions of EQ-5D-Y and EQ-HWB-S (EuroQol health and well-being questionnaire, short version), the study evaluates HRQoL changes over 1 and 2 years and explores the impact on caregiver burden and spillover effects. A control group of 100 healthy children and their parents will be included. Data collection involves baseline and follow-up surveys, clinical data from medical records, and statistical analyses to compare treatment effects and validate measurement tools.

DETAILED DESCRIPTION:
[Research Background] Asthma and allergic rhinitis are common chronic diseases in children, significantly impacting their HRQoL and increasing healthcare burden. Allergen-specific immunotherapy (AIT) is an effective treatment for these conditions, shown to improve symptoms and QoL. This study aims to further understand the impact of AIT on QoL in children and their caregivers, using validated assessment tools and comprehensive clinical data. The findings will contribute to better clinical management and policy-making for pediatric allergic diseases.

[Study Design] Prospective observational study.

[Primary Objectives] Assess the current health-related quality of life (HRQoL) of children with airway allergic diseases (bronchial asthma, allergic rhinitis, or both) using the EQ-5D-Y and disease-specific scales.

Evaluate and compare the dynamic changes in HRQoL over 1 and 2 years in children undergoing routine treatment versus specific immunotherapy. Analyze the impact of treatment type, disease severity, and treatment outcomes.

Determine the impact of allergic diseases on children's HRQoL by comparing them with healthy controls.

[Secondary Objectives] Explore the caregiver burden and spillover effects on parents using the PedsQL Family Impact Module, compared with healthy controls.

Compare the QoL of parents based on different treatment plans, disease severities, and treatment outcomes of their children.

Validate the newly developed Chinese versions of EQ-5D-Y and EQ-HWB-S for parents' QoL assessment.

[Participants] 200 children (ages 5-16) diagnosed with bronchial asthma, allergic rhinitis, or both, and their 200 parents (caregivers), divided into two groups: 100 children receiving specific immunotherapy and 100 receiving routine treatment.

Control group: 100 healthy children and their parents.

[Methods] Children with Allergies: Complete baseline and two follow-up surveys. Use the EQ-5D-Y-3L (3 level of EQ-5D-Y), EQ VAS (Visual Analogue Scale), PAQLQ (Pediatric Asthma Quality of Life Questionnaire) or JRQLQ-No. 1 (Japanese Rhinoconjunctivitis Quality of Life Questionnaire No. 1 ), and Overall Health Assessment (OHA).

Healthy Children: Complete a single baseline survey using EQ-5D-Y-3L, EQ VAS, and OHA.

Parents: Complete EQ-HWB-S, demographic information, EQ-5D-5L, OHA, and PedsQL (Pediatric Quality of Life Inventory) Family Impact Module.

Clinical data collection from medical records including diagnosis, symptoms, laboratory tests (lung function, allergens, eosinophils, IgE, FeNO[Fractional Exhaled Nitric Oxide]), treatment plans, side effects, and complications.

[Inclusion Criteria] Children with Allergies: Ages 5-16, diagnosed with bronchial asthma, allergic rhinitis, or both, with continuous treatment for ≥4 weeks. Able to understand and complete questionnaires.

Healthy Children: Ages 5-16, without a history of allergic diseases. Able to understand and complete questionnaires.

Parents: Primary caregivers, present during survey, signed informed consent.

[Study Endpoints] Completion of the second follow-up survey by the last enrolled child and parent.

[Primary Outcomes] Disease severity (Asthma Control Test, ACT). Laboratory tests (lung function, serum allergens, eosinophils, IgE, oral/nasal FeNO)

[Statistical Methods] Compare HRQoL before and after treatment in children and parents, and between allergic and healthy groups using t-tests, Wilcoxon rank-sum tests, chi-square tests, or Fisher's exact tests. Use ANOVA, Kruskal-Wallis tests, and chi-square tests for multiple group comparisons. Analyze correlations between HRQoL and influencing factors using multiple regression. Validate HRQoL scales using variance analysis for construct validity and effect size for responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Children:

   1. Aged 5-16 years;
   2. Diagnosed with bronchial asthma, allergic rhinitis, or both (persistent, duration ≥4 weeks) by a respiratory or allergy specialist;
   3. Guardian has signed the informed consent form;
   4. Able to understand and complete the questionnaire;
   5. Outpatients or inpatients at the Pediatrics Department of Renji Hospital in Shanghai.
2. Parents:

   1. The primary caregiver of the enrolled child;
   2. Accompanied the child to the hospital on the day of the visit;
   3. Signed the informed consent form;
   4. Able to understand and complete the questionnaire.

Exclusion Criteria:

1. Children:

   1. Poor compliance;
   2. Already received specific immunotherapy at another hospital;
   3. Unable to independently read and complete the questionnaire;
   4. Lost to follow-up or discontinued treatment.
2. Parents:

   1. Unwilling to sign the informed consent form;
   2. Unable to complete the questionnaire due to physical condition or educational level.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study involves 200 children aged 5-16 years diagnosed with bronchial asthma, allergic rhinitis, or both, along with their 200 parents (direct caregivers). Of these children, 100 will receive allergen-specific immunotherapy, while the other 100 will undergo conventional treatment. Additionally, the control group consists of 100 pairs of healthy children and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Asthma control level for asthmatic children | Baseline 1 week before treatment; 2 follow-up every 12 months
  The child or their parent recalls the frequency of asthma symptoms over the past four weeks, including daily activities, coughing, wheezing, use of asthma medications, and nighttime sleep. The attending physician collects this information during the consultation and assesses the severity of the condition. For individuals aged 12 and above, the Asthma Control Test (ACT) scores are interpreted as follows: a score of 25 or above indicates fully controlled asthma, 20-24 indicates well-controlled asthma, and 19 or below indicates uncontrolled asthma. For children aged 4 to 11, the Childhood Asthma Control Test (C-ACT) scores are interpreted similarly: a score of 24 or above indicates fully controlled asthma, 20-23 indicates well-controlled asthma, and 19 or below indicates uncontrolled asthma.
Severity assessment of allergic rhinitis | Baseline 1 week before treatment; 2 follow-up every 12 months
  The attending physician collects information on the patient's symptoms over the past four weeks, including sleep disturbances, limitations in daily activities such as leisure and exercise, limitations in learning, and symptoms (such as nasal itching, nasal congestion, runny nose, and sneezing) that did not cause significant discomfort. The physician then assesses the severity of the condition based on this information. Mild: None of the following are present: sleep disturbances, limitations on daily activities such as leisure/sports, learning limitations, and symptoms (itchy nose, nasal congestion, runny nose, sneezing) that do not cause distress. Moderate to Severe: One or more of the above symptoms are present.
EQ-5D-Y-3L for assessing health-related quality of life | Baseline 1 week before treatment; 2 follow-up every 12 months
  The EQ-5D-Y-3L assesses HRQoL with five dimensions (mobility; looking after myself; doing usual activities; having pain or discomfort; and feeling worried, sad, or unhappy) and three severity levels. Each health state in the EQ-5D-Y-3L can be summarized using level descriptors, generating 243 (35) unique states. The best state, 11111, indicates 'no problems' in any dimension, while the worst state, 33333, indicates 'a lot of problems' in all dimensions. An index score of 1.0 represent the value of full health, and a score of 0.0 the value of death. Negative values represent health states with values below the value of death.
EQ-VAS for assessing health-related quality of life | Baseline 1 week before treatment; 2 follow-up every 12 months
  A 20-cm visual analogue scale for overall health rating. Higher indicates better HRQoL.
PAQLQ for assessing health-related quality of life in children with asthma | Baseline 1 week before treatment; 2 follow-up every 12 months
  The questionnaire includes symptoms (10 questions), activities (5 questions), and emotional functioning (8 questions), using a 7-point scale where 1 is the worst and 7 is the best. The total score is the sum of the scores for each dimension, with higher scores indicating better quality of life and lower scores indicating worse quality of life. A score greater than 66% of the total possible score indicates a high quality of life, 33%-66% indicates a moderate quality of life, and less than 33% indicates a low quality of life.
JRQLQ-No. 1 for assessing health-related quality of life in children with allergic rhinitis | Baseline 1 week before treatment; 2 follow-up every 12 months
  The JRQLQ-No.1 questionnaire consists of 3 sections with a total of 24 items. Scoring: Calculate the average score for the first and second sections, then add the scores of all three sections and calculate the overall average score. Each item is scored on a scale, where higher scores indicate a better quality of life and lower scores indicate a worse quality of life. The minimum possible score is 1, indicating the worst outcome, and the maximum possible score is 7, indicating the best outcome.

SECONDARY OUTCOMES:
Pulmonary function for assessing asthma disease severity | Baseline 1 week before treatment; 2 follow-up every 12 months
  Pulmonary function tests include various measurements to assess lung function. Vital capacity measurement determines the maximum amount of air a person can exhale after a maximum inhalation, which helps diagnose conditions like restrictive lung disease. Peak expiratory flow rate (PEFR) measures the highest speed of exhalation, useful in evaluating airway obstruction, commonly in asthma management. Lung volumes include measurements of different capacities, such as total lung capacity, providing insights into lung function. Additionally, diffusion capacity tests assess how well gases like oxygen move from the lungs into the blood, crucial for identifying issues like pulmonary fibrosis or emphysema. PEFR and FEV1 values within 80-100% of the predicted range and a normal FEV1/FVC ratio indicate well-controlled asthma and normal lung function.
Peripheral Blood Eosinophils for assessing allergic severity | Baseline 1 week before treatment; 2 follow-up every 12 months
  Peripheral blood eosinophil counts are used to assess the severity of allergic conditions. Normal levels are less than 500 eosinophils per microliter of blood. Elevated counts (eosinophilia) indicate allergic reactions or conditions such as asthma, allergic rhinitis, chronic rhinosinusitis with nasal polyps, and eosinophilic esophagitis. Higher eosinophil levels can help in diagnosing allergies, monitoring treatment effectiveness, predicting exacerbations, and guiding the use of biologic therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjing Zhou, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided